CLINICAL TRIAL: NCT06399601
Title: A Training Program of Drug Allergy for Healthcare Professionals: A Randomized Controlled Trial
Brief Title: A Training Program of Drug Allergy for Healthcare Professionals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Drugallergy
Record Dates: First submitted 2024-04-09; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Drug Allergy
Keywords: Drug allergy
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): wo identical didactic courses on drug allergy will be delivered. Changes in knowledge and clinical practice will be measured by serial practice questionnaires and knowledge quizzes conducted before and after the course. Group 1 will undergo the course first.
  Interventions: Other: Drug allergy training program
- Control group (Active Comparator): Group 2 will undergo an identical course one month later. By comparing any changes in knowledge or practice between groups, this ensures that any changes in knowledge or practice were solely due to the course and not other external factors.
  Interventions: Other: Drug allergy training program

INTERVENTIONS:
Other: Drug allergy training program — Two identical didactic courses on drug allergy were designed. Each course will last 12 hours and conducted over 2 consecutive days (6 hours each day). All candidates will attend physically and on-site. Various aspects of drug allergy with pre-set learning objectives will be taught in-person by instructors (physicians or nurses specializing in drug allergy nominated by the University of Hong Kong). Course materials and instructors will be identical for each course.

SUMMARY:
Drug allergy is often under-recognized, yet over- (mistakenly) diagnosed, especially in Hong Kong. There is also a dire shortage of allergy specialists and facilities to tackle the overwhelming drug allergy pandemic. Fortunately, when trained, non-specialist physicians and nurses have demonstrated comparable capabilities in drug allergy evaluation compared to specialists. To potentially promote and propagate the role of non-specialist physicians and nurses toward drug allergy care, the investigators propose a study to investigate the impact of an intensive and focused drug allergy educational course conducted at the University of Hong Kong.

DETAILED DESCRIPTION:
Two identical didactic courses on drug allergy were designed. Each course will last 12 hours and conducted over 2 consecutive days (6 hours each day). All candidates will attend physically and on-site. Various aspects of drug allergy with pre-set learning objectives will be taught in-person by instructors (physicians or nurses specializing in drug allergy nominated by the University of Hong Kong). Course materials and instructors will be identical for each course.

Aims of the study Primary objective

* Investigate the change in knowledge among participants of a 2-day drug allergy educational course
* Investigate the change in clinical practice among participants of a 2-day drug allergy educational course

Secondary objectives

* Investigate the sustained change(s) in knowledge (if any) of participants of a 2-day drug allergy educational course
* Investigate the sustained change(s) in clinical practice (if any) of participants of a 2-day drug allergy educational course

Hypothesis The investigators hypothesize that candidates (practicing physicians and nurses) of the drug allergy course will gain knowledge on drug allergy, which in turn will influence and change their clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses or doctors actively practicing in Hong Kong
* English speaking;
* Able to complete quizzes and questionnaires;
* Aged 18 or above

Exclusion Criteria:

* People who are unable to communicate in Cantonese or Mandarin
* People who are participating in other drug allergy training course

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge of drug allergy as measured by the validated drug allergy questionnaire | After the 2-day training course
  Knowledge includes mechanism, clinical manifestations, diagnosis and management of drug allergy. A binary variable scale were used to ascertain level of the knowledge (from 0 to 1: 0, wrong; 1, right). Answers formats consisted of 4-choice questions (total 14 questions).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Biomedical Science, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mak HWF, Meng J, Chung FKL, Lee JTY, Aberathna IS, Amarasekara U, Ranasinghe TND, Jayamali J, Yang Q, Zhou M, Chen L, Huang JX, Shi W, Kulkarni R, Peter JG, Trubiano JA, Jeewandara KC, Lucas M, Li PH. Bridging Global Disparities in Drug Allergy Through AI-Assisted Training for Non-Specialists: Findings From the Multinational ADAPT-2 Course. Clin Exp Allergy. 2026 Jan 20. doi: 10.1111/cea.70213. Online ahead of print. PMID 41558734